CLINICAL TRIAL: NCT03304886
Title: Diagnostic Comparison of an Online Questionnaire Versus a Semi-structured Interview for the Diagnosis of Primary Headache Disorders, Using ICHD 3 as the Gold Standard
Brief Title: Assessing the Diagnostic Accuracy of an On-line Questionnaire for Diagnosis of Primary Headache Disorders
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Cowan, Director and Chief, Division of Headache Medicine, Stanford University
Other Study IDs: John Henry study
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraineurs: with a migraine
- Control: Participants without migraine

SUMMARY:
Purpose of the study is to assess the diagnostic accuracy of an on- line questionnaire in comparison to a semi-structured interview administered by a trained interviewer.

DETAILED DESCRIPTION:
The worldwide current gold standard for diagnosing headaches is the International Classification of Headache Disorders (ICHD 3 beta). Adhering strictly to ICHD criteria has been problematic for accurately diagnosing patients in the clinic and as for clinical trials. To address these issues, an online instrument was developed that successfully diagnosis common primary and secondary headache disorders. In this research Investigator hopes to demonstrate an on- line questionnaire is non inferior to a semi-structured interview for accurately diagnosing different types of headaches (for example: episodic migraine vs. non episodic migraine, chronic migraine vs. non chronic migraine, episodic tension-type vs. non-episodic tension type, chronic tension-type headache vs. non chronic tension-type headache, medication overuse headache vs. non medication overuse headache, post traumatic headache vs. non post traumatic headache).

Participants will be screened by telephone to see if participants meet the criteria for taking part in this research study. Once participant is deemed eligible,the participants will then be randomized in a 1:1 ratio to complete either the semi-structured interview over the phone first and then complete the online questionnaire or vice versa. Study is expected to enroll 500 participants with headache and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects age between age 18-65(inclusive),
2. Subjects must agree to sign online informed consent;
3. Subject must be able to understand and willing to complete both evaluations in English
4. Willing to comply with study instructions.
5. Agree not to Rely or act on any diagnosis given to them in the study

Exclusion Criteria:

1. Presence of Disorders listed in groups 5-13 of The International Headache Society Classification of Head and Facial Pain (Headache Classification Committee of the International Headache Society, 2015 except for post traumatic headache and medication overuse headache);

1a. History of brain tumor, brain surgery

1b. History of brain infection such as meningitis, encephalitis, or meningoencephalitis

1c. History of any significant current or previous brain dysfunction

1d. Regular use of illicit drugs.

2. Known significant medical or psychiatric disease or abnormal laboratory data that would preclude entry into this study.

3. Subjects with - significant cognitive impairment such as dementia, active psychiatric disease such as schizophrenia.

4. Subjects with physical limitations to participate in the on-line or phone interview impossible.

5. Non-English speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All race, gender age between 18-65, English speaking selected from community, clinic.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
On-line questionnaire accuracy for Diagnosing episodic migraine | 2 -2.5 years
  An on- line questionnaire is non inferior to a semi-structured interview for accurately diagnosing episodic migraine vs non episodic migraine, chronic migraine vs. non chronic migraine. We will compare the 4 primary (chronic and episodic migraine, chronic and episodic tension-type headache) obtained on each of the two evaluations for reliability using recognized statistical tools: This analysis will be conducted by independent reviewers, not the developers of either instrument

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, MD, FAAN, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeSouza DD, Woldeamanuel YW, Sanjanwala BM, Bissell DA, Bishop JH, Peretz A, Cowan RP. Altered structural brain network topology in chronic migraine. Brain Struct Funct. 2020 Jan;225(1):161-172. doi: 10.1007/s00429-019-01994-7. Epub 2019 Dec 2. PMID 31792696